CLINICAL TRIAL: NCT02473913
Title: Silymarin Treatment of Trichotillomania in Children and Adults: A Double-Blind, Placebo-Controlled, Cross-Over Study
Brief Title: Milk Thistle in Trichotillomania in Children and Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0178
Record Dates: First submitted 2015-06-02; First posted 2015-06-17 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Trichotillomania; Hair Pulling Disorder
MeSH Terms: conditions — Trichotillomania | interventions — milk-thistle extract; Silymarin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milk Thistle (Experimental): Each subject will have a 6 week treatment phase with milk thistle.
  Interventions: Drug: Milk Thistle
- Placebo (Placebo Comparator): 6 week placebo phase before or after milk thistle phase depending on randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milk Thistle
  Other Names: Silymarin
  Arms: Milk Thistle
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of silymarin (milk thistle) in children and adults with trichotillomania. The hypothesis to be tested is that silymarin will be more effective and well tolerated in children and adults with trichotillomania compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
Pathological hair-pulling, trichotillomania, has been defined as repetitive, intentionally performed pulling that causes noticeable hair loss and results in clinically significant distress or functional impairment. Trichotillomania appears relatively common with an estimated prevalence between 1-3%. Data on the pharmacological treatment of trichotillomania is limited to case reports and conflicting double-blind studies of serotonin reuptake inhibitors. One positive double-blind study of N-acetyl cysteine in adults was not successful when examined for children and adolescents. Available data on the treatment of trichotillomania in children are therefore limited.

Silymarin, a flavonoid and a member of the Asteraceae family, is extracted from the seeds of milk thistle (Silybum marianum) and is known to have antioxidative and anti-apoptotic properties. Furthermore, it has been demonstrated that its anti-oxidative activity is related to the scavenging of free radicals and activation of anti-oxidative defenses: increases in cellular glutathione content and superoxide dismutase activity. Milk thistle has been used for a range of psychiatric disorders including methamphetamine abuse and obsessive compulsive disorder. The flavonoid complex silymarin in preclinical studies has been found to increase serotonin and dopamine levels in the cortex. In the frontal cortex one of the functions of dopamine is to increase the signal to noise ratio, increased dopamine correlating with increased frontal performance. Studies have shown that the higher cortical dopamine levels are associated with improved frontal cortical cognitive performance. Cortical inhibition is felt to be the basis for top-down control of motivated behaviors. A recent randomized controlled study with milk thistle was conducted in Iran Thirty five participants with moderate OCD were randomly assigned to 200 mg of milk thistle leaf extract or 10 mg of fluoxetine three times daily for eight weeks. Results revealed no significant difference in treatment effects between milk thistle and fluoxetine from baseline to endpoint as both interventions provided a highly significant reduction in symptoms. Silymarin or Milk Thistle may therefore offer promise for the treatment of individuals with trichotillomania.

The current pilot study examines the tolerability and efficacy of milk thistle in the treatment of trichotillomania in children and adults. The investigators hypothesize that milk thistle will reduce the severity of symptoms related to trichotillomania and improve patients' overall functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 10-65.
2. Diagnosis of current trichotillomania (TTM) based on DSM-5 criteria and confirmed using the clinician-administered Structured Clinical Interview for DSM-5 (SCID);
3. Hair-pulling behavior within 2 weeks prior to enrollment;
4. Child able and willing to provide active assent for participation;
5. Legal guardian available to provide consent for participation.

Exclusion Criteria:

1. Infrequent hair-pulling (i.e. less than one time per week) that does not meet DSM-5 criteria for trichotillomania;
2. Unstable medical illness as determined by the investigator;
3. History of seizures;
4. Current use of stimulants coinciding with onset or exacerbation of trichotillomania symptoms or other current medications coinciding with exacerbation or onset or trichotillomania symptoms;
5. Clinically significant suicidality (defined by the Columbia Suicide Severity Rating Scale);
6. Baseline score of ≥17 on the Hamilton Depression Rating Scale (17-item HDRS);
7. Lifetime history of bipolar disorder type I or II, schizophrenia, autism, any psychotic disorder, or any substance use disorder;
8. Initiation of psychotherapy or behavior therapy within 3 months prior to study baseline;
9. Previous treatment with milk thistle;
10. Any history of psychiatric hospitalization in the past year.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-03; Primary Completion 2018-06 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover study. Therefore, only 22 participants were technically enrolled, but they each were supposed to complete both the placebo and the Milk Thistle Arm.
Groups:
- Experimental: Milk Thistle, Then Placebo: Participants first received Milk Thistle for 6 weeks. After a washout period of 1 week, they then received matching Placebo for 6 weeks.
- Experimetal: Placebo, Then Milk Thistle: Participants first received matching Placebo for 6 weeks. After a washout period of 1 week, they then received matching Milk Thistle for 6 weeks.
Period: Overall Study
Arm/Group | Experimental: Milk Thistle, Then Placebo | Experimetal: Placebo, Then Milk Thistle
Started | 11 | 11
Completed | 8 | 8
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Milk Thistle, Then Placebo: Participants first received Milk Thistle for 6 weeks. After a washout period of 1 week, they then received matching placebo for 6 weeks.
- Placebo, Then Milk Thistle: Participants first received matching placebo for 6 weeks. After a washout period of 1 week, they then received Milk Thistle for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Milk Thistle, Then Placebo | Placebo, Then Milk Thistle | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (11.5) | 27.7 (11.1) | 28.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 7 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in NIMH Trichotillomania Severity Scale (NIMH-TSS) Scores
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the NIMH-Trichotillomania Symptom Severity Scale (NIMH-TSS). The change in scores from baseline to after 13 weeks will be assessed. The NIMH-TSS consists of 5 questions related to the following aspects of TTM: average time spent pulling, time spent pulling on the previous day, resistance to urges, resulting distress and daily interference. NIMH-TSS scores range from 0 to 25, with higher scores indicating higher severity.
Time Frame: Baseline and 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Milk Thistle: Each subject will have a 6 week treatment phase with milk thistle.
  Milk Thistle
- Placebo: 6 week placebo phase before or after milk thistle phase depending on randomization.
  Placebo
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-Treatment | 9.4 (5.4) | 9.4 (5.0)
  Post-Treatment | 6.3 (5.3) | 7.4 (5.1)

2. Secondary Outcome: Massachusetts General Hospital Hair Pulling Scale (MGH-HPS)
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the MGH-Hair Pulling Scale (MGH-HPS). At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported. The MGH-HPS is a self report scale that assesses severity of Trichotillomania in the past week. There are seven total items each rated for severity from 0 to 4. Higher scores indicate higher symptom severity.
Time Frame: Up to 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-Treatment | 13.5 (6.8) | 14.7 (7.1)
  Post-Treatment | 10.4 (7.6) | 12.3 (6.5)

3. Secondary Outcome: Clinical Global Impression- Severity and Improvement (CGI)
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the CGI. At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported. The CGI-Severity is rated on a 7-point scale, with the severity of illness ranging from 1 (normal) through 7 (among the most severely ill patients). CGI-Change scores range from 1 (very much improved) through 7 (very much worse).
Time Frame: Up to 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Pre-Treatment | 4.1 (1.0) | 3.9 (0.6)
  Post-Treatment | 3.0 (1.4) | 3.6 (0.9)

4. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the Sheehan Disability Scale (SDS). At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported. The scale itself assesses the level of functional impairment from trichotillomania (or target disorder). The subject is asked to rank the extent to which work/school, family life/home responsibilities, or social life are impaired by their symptoms on a scale from 0 (not at all) to 10 (extremely). The three numerical ratings can then be summed to produce a single measure of global functional impairment from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Up to 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-Treatment | 8.8 (8.0) | 8.8 (4.1)
  Post-Treatment | 5.2 (7.8) | 5.9 (7.1)

5. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the Hamilton Anxiety Rating Scale (HAM-A), a 14 item scale. At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Up to 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-Treatment | 4.9 (4.8) | 5.1 (4.4)
  Post-Treatment | 2.8 (3.5) | 3.4 (3.0)

6. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The entire study for the subject will last 13 weeks. Every two weeks and after the one week washout period the subject will take the Hamilton Depression Rating Scale (HAM-D). At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported.
  Classification of symptoms are scored as follows:
  0 - absent: 1 - doubtful or trivial: 2 - present.
  Classification of symptoms where more detail can be obtained can be expanded to:
  0 - absent; 1 - mild; 2 - moderate; 3 - severe; 4 - incapacitating.
  In general the higher the total score the more severe the depression. HAM-D score level of depression:
  10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Time Frame: Up to 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-Treatment | 5.7 (5.1) | 5.5 (4.4)
  Post-Treatment | 2.7 (3.3) | 2.9 (3.1)

7. Secondary Outcome: Trichotillomania Scale for Children/Parent (TSC-C & TSC-P)
Description: The entire study for the subject will last 13 weeks. The subject will take the TSC-C (child version).The parent of the subject will fill out the TSC-P (parent version). At each of these visits the outcome will be assessed. Pre treatment and after the one week washout period scores reported. The scale itself assesses severity of trichotillomania and provides a sub score for severity. The severity score is produced by adding up the scores for questions 1 through 5 and dividing that sum by 5. The second sub score is on distress/impairment with questions such as "in the past week, how often did you feel like pulling your hair?". The sub score for distress/impairment is produced by adding the scores for questions 6-12 and dividing that sum by 7. The sum of both sub scores provides a total score. Total scores (ranging between 0 and 4) were compared pre treatment and post treatment. Higher scores indicate a higher severity and distress impairment score.
Time Frame: Up to 13 weeks
Population: For some subjects, the scale was not filled out at follow-up visits (in error).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milk Thistle | Placebo
Number analyzed (Participants) | 3 | 3
score on a scale
  Pre-Treatment (TSC-C) | 2.9 (0.3) | 2.0 (0.8)
  Post-Treatment (TSC-C): number analyzed (Participants) | 3 | 2
  Post-Treatment (TSC-C) | 1.7 (1.1) | 1.7 (0.1)
  Pre-Treatment (TSC-P) | 2.5 (0.2) | 1.9 (0.1)
  Post-Treatment (TSC-P): number analyzed (Participants) | 2 | 2
  Post-Treatment (TSC-P) | 1.1 (0) | 2.3 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each study visit (Visits 1-8) over the subjects' study participation (13 weeks) and over the total course of the study (3 years).
Arm/Group | Milk Thistle | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 6/18 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milk Thistle (N=18) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT02473913/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02473913/ICF_001.pdf